CLINICAL TRIAL: NCT07389707
Title: The Effect of Using Hand Massage Stimulation Techniques on Pain and Comfort in Pregnant Women Experiencing Lumbar Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra Tan, master thesis student, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/129
Record Dates: First submitted 2026-01-27; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Related
Keywords: back pain; comfort; pregnant; massage; midwife
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Crossover Assignment randomized controlled trial conducted with experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- seed therapy ( su-jok) (Experimental): Group that received seed therapy ( su- jok )
  Interventions: Other: seed therapy (su-jok)
- standard maintenance (No Intervention): group not receiving seed therapy ( su- jok)

INTERVENTIONS:
Other: seed therapy (su-jok) — In hand massage, tiny swellings called "ball conformity" occur on the reflection points of the organs where the complaint occurs on the hands and feet. It is argued that the sensitivity of the relevant point to pressure has a direct correlation with the level of pain in the body part. A rod called a "diagnostic probe" or "diagnostic rod" made of metal, plastic or wood, approximately ten centimeters long, is used to detect the painful point on the hand and foot. After the correct point is detected, various techniques are applied to stimulate these points and ensure the continuation of the energy flow.In this study, the seed massage technique, which does not cause any side effects among the hand massage stimulation methods, requires a basic level certificate for its use, does not require being a health professional, and can be easily applied by anyone, will be used. Seed massage is a method applied by first detecting pain through a probe on the points of the organs reflected on the hand
  Arms: seed therapy ( su-jok)

SUMMARY:
The aim of this study is to determine the effects of hand massage stimulation techniques applied to pregnant women with low back pain on pain and comfort.

H1-a: Hand massage stimulation technique applied to pregnant women reduces low back pain.

H1-b: Hand massage stimulation technique applied to pregnant women increases comfort Data will be collected from pregnant women who apply to the NST polyclinic and complain of back pain. Midwifery intervention will be implemented in a way that does not disrupt the examination routine. Seed therapy (su-jok) will be applied by researcher Esra Tan, who has a basic level su jok therapy certificate.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of hand massage stimulation techniques applied to pregnant women with low back pain on pain and comfort.

Data will be collected from pregnant women who apply to the NST polyclinic in the gynecology and obstetrics clinic of the Adıyaman Gölbaşı State Hospital and complain of back pain. Participants who meet the inclusion criteria and agree to participate will be informed about the study and participants who fill out the "Minimum Informed Consent Form" will be included in the study. Data collection forms will be applied by the researcher, paying attention to patient privacy, and the pre-test data collection phase will be completed. After the pre-test data collection phase is completed, hand stimulation techniques (su-jok seed therapy) will be applied to the pregnant women in the experimental group by the researcher. Pregnant women will be invited to the pregnancy education class in the relevant hospital and detailed information will be given about the application, and pain points will be determined according to the reflections of the organs on the hand. Buckwheat seeds, one of the seeds used for back pain, will be fixed on the detected points and the fixed seed will be removed after 5-6 hours. This application will be done in 1 session and the post-test will be applied 15 minutes after the seed is removed. This intervention will be implemented by Esra Tan and the researcher has a basic level su jok therapy certificate. No intervention will be applied to the pregnant women in the control group, however, the Personal Information Form, Visual Analog Scale (VAS), Prenatal Comfort Scale and Oswestry Disability Index will be applied simultaneously with the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are over 18 years old,
* Able to read and write,
* Have back pain severity of 45 mm and above according to Visual Analogue Scale (VAS),
* Aren't experiencing risky pregnancies,
* Do not have any psychiatric disorders,
* Have a gestational age of 32 weeks or above,
* Do not react negatively to any interventions such as massage,
* Have healthy and complete tissue integrity in the area where the massage will be performed will be included in the sample.

Exclusion Criteria:

* Pregnant women with acute or chronic diseases, traumas, or surgical history related to the musculoskeletal or nervous system,
* Those who have gynecological or urological problems that cause pain during pregnancy (premature birth, pyelonephritis, etc.),
* Those who use analgesics during pregnancy,
* Those who have difficulty communicating and mentally ill,
* Those who have a condition that may prevent written or verbal communication,
* Those who have maternal and fetal complications in their current pregnancy will not be included in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Prenatal Comfort Scale scores | At baseline (pre-intervention) and immediately after completion of seed therapy]
  The initial version of the scale consisted of 34 items, but was later revised by the authors and shortened to 15 items (21). The short version of the scale consists of 15 items and 5 sub-dimensions. Each item is scored between 0-5 (0=Strongly disagree, 1=Disagree, 2=Undecided, 3=Somewhat agree, 4=Agree, 5=Strongly agree). The scale is evaluated out of a total of 75 points.

SECONDARY OUTCOMES:
Oswestry Disability Index scores | At baseline (pre-intervention) and immediately after completion of seed therapy
  It consists of 10 questions, each scored between 0 and 5, that examine the severity of pain, personal care, lifting, walking, sitting, standing, sleeping, social life, travel and the degree of change in pain in order to evaluate the effect of low back pain on daily activities. The quality of life increases as the score obtained from the Oswestry Disability Index decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Esra GÜNEY, PhD, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Battalgazi̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared

REFERENCES:
- See also: Reference link — https://pubmed.ncbi.nlm.nih.gov/39561422/